CLINICAL TRIAL: NCT05551780
Title: Treatment of Calcific Total Occlusions in Peripheral Artery Disease
Acronym: CaTO-PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SoundBite Medical Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT-PER-2022-01
Record Dates: First submitted 2022-09-14; First posted 2022-09-23 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Chronic Total Occlusion of Artery of the Extremities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SoundBite Crossing System - PAD (Experimental): Use of the SoundBite Crossing System to cross calcified chronic total occlusions (above-the-knee or below-the-knee)
  Interventions: Device: SoundBite Crossing System
- SoundBite Crossing System - BTK (Experimental): Use of the SoundBite Crossing System to cross calcified chronic total occlusions (below-the-knee)
  Interventions: Device: SoundBite Crossing System

INTERVENTIONS:
Device: SoundBite Crossing System — Use of the SoundBite Crossing System to cross calcified chronic total occlusions

SUMMARY:
Prospective, multi-center, non-randomized, open label, clinical study intended to provide data to demonstrate safety and performance of the SoundBite Crossing System XS Peripheral.

DETAILED DESCRIPTION:
The CaTO-PAD study includes a below-the-knee (BTK) sub-study (CaTO-BTK)

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for interventional treatment of de-novo lesion(s) of the following native arteries:

   1. CaTO-PAD: infrainguinal
   2. CaTO-BTK: infrapopliteal
2. Have at least one chronic total occlusion (CTO) with no flow observed in the distal lesion except the flow from collateral circulation
3. Presenting with the following:

   1. CaTO-PAD: claudication or CLI (Rutherford Clinical Category 2-5) of the target limb
   2. CaTO-BTK Sub-Study: - Category 4 or 5 only for CaTO-BTK Sub-Study CaTO-PAD: claudication or CLI (Rutherford Clinical Category 2-5) of the target limb
4. Age of > 18 years
5. Have been informed of the nature of the study, agrees to participate, and has signed the approved study consent form
6. Target lesion calcification is at least moderate by PARC definition (see Section 15)
7. Target lesion is refractory as demonstrated by a failed attempt with a guidewire

Exclusion Criteria:

1. Any medical condition that would make subject an inappropriate candidate for interventional treatment as determined by the Investigator, including the following:

   1. Glomerular filtration rate <30 ml/min
   2. Mortality expected within 30 days
2. Already enrolled in an investigational interventional study that would interfere with study endpoints
3. Target lesion is crossed intraluminally with a conventional guidewire
4. Treatment of an inflow lesion prior to target lesion treatment results in no reflow, thrombus formation, abrupt closure, distal embolization, dissection or perforation requiring treatment
5. Women who are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Device Performance | Day 0
  Crossing of the lesion regardless of method or modality (e.g., antegrade or retrograde)
Device Safety | Day 0
  Procedural incidence of any of the following: no reflow, thrombus formation, abrupt closure, distal embolization, dissection or perforation requiring treatment

SECONDARY OUTCOMES:
Antegrade Crossing | Day 0
  Placement of a guidewire distal to the lesion in the true lumen (Note: retrograde crossing is allowed, but is considered a failure for this endpoint)
CTO Crossing Time | Day 0
  From first engagement of proximal cap with the Active Wire to guidewire in distal true lumen (or decision made to discontinue attempts)
Acute Lumen Gain | Day 0
  Difference in final minimal lumen diameter compared to baseline
Residual Percent Stenosis | Day 0
  Final percent stenosis at procedure end
Procedure Time | Day 0
  First groin puncture to final sheath removal
Fluoroscopy Time | Day 0
Number of Devices Used | Day 0
  Conventional guidewires, microcatheters, atherectomy devices, re-entry devices, balloons, stents
Secondary Safety Endpoint | Day 30 (+10/-0 days)
  Rate of 30-day major adverse events (MAE) consisting of: death, emergency surgical revascularization of the target limb, unplanned amputation of the target limb, symptomatic distal thrombus or emboli requiring intervention, perforation requiring treatment

CONTACTS AND LOCATIONS:
Overall Officials: George Adams, MD, Principal Investigator — UNC REX Hospital, Raleigh, NC, USA; Michael Lichtenberg, MD, Principal Investigator — Angiology Clinic and Vascular Centre, Arnsberg, Germany
Locations (5):
- United States (3):
  - Palm Vascular Centers, Fort Lauderdale, Florida
  - UNC REX Hospial, Raleigh, North Carolina
  - Lifespan - The Miriam Hospital, Providence, Rhode Island
- Medizinische Universität Graz, Graz, Austria
- Angiology Clinic and Vascular Centre, Arnsberg, Germany

IPD SHARING:
Plan to Share IPD: No